CLINICAL TRIAL: NCT04138602
Title: A Single-Blind, Randomized, Pilot Study of the BTL Emsella Chair With Dietary Counseling Versus Sham Chair With Dietary Counseling for the Treatment of Fecal Incontinence
Brief Title: BTL Emsella Chair Versus Sham for the Treatment of Fecal Incontinence
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kenneth M Peters, MD, Director and Chair of the Department of Urology, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-305
Record Dates: First submitted 2019-10-16; First posted 2019-10-24 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Fecal Incontinence
Keywords: Fecal smearing; Incomplete defecation; Fecal urgency
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: Patients who meet all the eligibility criteria will be enrolled in the study and randomized (1:1) to receive Emsella Chair or sham treatments. Randomization will be performed using a table of random numbers. Randomization envelopes will be provided by the study's biostatistician and will be securely stored in a locked cabinet. The study coordinator(s) will solely be responsible for opening the randomization envelopes and delivering the study treatments, according to the group assignment. Ultimately, they will be responsible for maintaining the confidentiality and security of the randomization envelopes. After the participant is randomized, the study coordinator(s) will complete the Subject Enrollment and Randomization Log. The log will be stored in the regulatory binder. The biostatistician will prepare more envelopes, if necessary.
  The patient will be given active Emsella treatment at the therapeutic level.
Who Masked: Participant
Masking Description: Patients who meet all the eligibility criteria will be enrolled in the study and randomized (1:1) to receive Emsella Chair or sham treatments. Randomization will be performed using a table of random numbers. Randomization envelopes will be provided by the study's biostatistician and will be securely stored in a locked cabinet. The study coordinator(s) will solely be responsible for opening the randomization envelopes and delivering the study treatments, according to the group assignment. Ultimately, they will be responsible for maintaining the confidentiality and security of the randomization envelopes. After the participant is randomized, the study coordinator(s) will complete the Subject Enrollment and Randomization Log. The log will be stored in the regulatory binder. The biostatistician will prepare more envelopes, if necessary.
  The sham Emsella treatment will provide sensation without active HIFEM technology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Emsella Chair Active Treatment with Dietary Counseling (Active Comparator): Subjects will be asked to sit on the device and the height will be adjusted until the subject's feet are on the floor. The active treatments are individualized, since some subjects will be more sensitive than others. The Emsella Chair will be turned on and the setting gradually increased to the subject's sensory threshold; the maximum sensation the subject can tolerate. The setting will then be decreased slightly and stay unchanged for the remainder of the treatment time. The treatment threshold should be increased with every treatment until the subject reaches 100%. During the visit the subject will also receive dietary counseling.
  Interventions: Device: BTL Emsella
- Emsella Sham Treatment with Dietary Counseling (Placebo Comparator): Sham subjects will be positioned on the device in the same manner. The sham treatment will provide some sensation without active HIFEM technology. The programming for the sham treatment will have an amplitude limitation, with the setting below therapeutic level (<10% power). During the visit the subject will also receive dietary counseling.
  Interventions: Device: Sham BTL Emsella

INTERVENTIONS:
Device: BTL Emsella — Subjects will be asked to sit on the device and the height will be adjusted until the subject's feet are on the floor. The active treatments are individualized, since some subjects will be more sensitive than others. The Emsella Chair will be turned on and the setting gradually increased to the subject's sensory threshold; the maximum sensation the subject can tolerate. The setting will then be decreased slightly and stay unchanged for the remainder of the treatment time. The treatment threshold should be increased with every treatment until the subject reaches 100%.
  Arms: Emsella Chair Active Treatment with Dietary Counseling
Device: Sham BTL Emsella — Sham subjects will be seated on the device in the same manner as the active treatment group. The sham treatment will provide some sensation without active HIFEM technology. The programming for the sham treatment will have an amplitude limitation, with the setting below the therapeutic level ( < 10 % power).
  Arms: Emsella Sham Treatment with Dietary Counseling

SUMMARY:
The purpose of this clinical trial is to compare the Emsella Chair to sham and to determine whether electromagnetic technology is effective in the treatment of fecal incontinence. Currently there are no other studies utilizing the Emsella Chair for the treatment of fecal incontinence. Eligible subjects will receive 2 treatments per week for a total of 4 weeks.

DETAILED DESCRIPTION:
Fecal incontinence, no matter how frequent, may significantly affect a patient's quality of life. Current available treatment options include; establishing a bowel regimen that consists of supplements, over the counter medications (stool softeners, laxatives, anti-diarrheal, enemas), or utilizing other prescription drugs (Linzees, Lomotil). Other conservative treatments include biofeedback therapy with a physical therapist. More invasive procedures include the injection of bulking agents or sacral nerve stimulation implantation.

The Emsella chair is currently approved as a treatment for stress urinary incontinence. The Emsella chair generates electromagnetic stimulation which is able to penetrate deep into the pelvic floor muscles inducing stimulation and providing rehabilitation for weak pelvic floor muscles. The Emsella Chair is a novel high-intensity focused electromagnetic (HIFEM) technology for the treatment of SUI, in addition to other pelvic floor related disorders. HIFEM technology induces deep pelvic floor muscle contractions designed to deliver the equivalent of 11,200 Kegel exercises over 28 minutes.

Subjects meeting eligibility will be randomized (1:1) to receive treatment with the Emsella chair and dietary counseling or sham Emsella chair with dietary counseling. A total of 8 treatments (2 treatments per week for 4 weeks) will be completed. For treatment delivery, participants will sit on the device and the chair height will be adjusted to ensure the subject's feet are on the floor. The sham Emsella treatment will provide some sensation without active HIFEM technology.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and provide written, dated, informed consent prior to screening, and be likely to comply with study protocol, including independently complete study questionnaires and communicate with study personnel about AEs and other clinically important information.
2. Women and men, 18 years of age or older
3. Subject reported fecal incontinence
4. Up to date on screening colonoscopy per guidelines (USPSTF)
5. Willingness to comply with conservative dietary management
6. Subject agrees to maintain a stable dose of any medication, prescribed or over the counter, known to affect bowel functioning.
7. Subject agrees not to start any new treatment (medication or otherwise) during the treatment and follow-up periods.
8. If of child-bearing age, agree to practice approved birth-control methods listed in appendix C

Exclusion Criteria:

1. Pregnant, or planning to become pregnant, at screening or anytime throughout the study period
2. Subject weighs more than 330 pounds
3. Pelvic floor physical therapy, including muscle training and/or electrostimulation, in a clinical setting within 30 days prior to screening
4. Pulmonary insufficiency, defined as difficulty breathing and fatigue, especially during exercise; chest pain, such as squeezing, pressure of tightness; the sensation of rapid or irregular heartbeat (palpitations); swelling of the legs or feet; dizziness or fainting; and/or bluish discoloration of the nails and/or lips (cyanosis)
5. Any condition that causes a lack of normal skin sensation to the pelvis, buttocks, and lower extremities
6. Major metal implants such as: metal plates, screws, joint replacements, implanted cardiac pacemakers, drug pumps, neurostimulators, electronic implants, copper intrauterine devices, defibrillators, and metal implants in the pelvic area. Patients with other metal implants will be evaluated by the investigator for inclusion in the study
7. Subject has a piercing between the waist and knees and is not willing to remove it before each treatment
8. Currently healing from surgical procedures where muscle contraction may disrupt the healing process
9. Subject has a malignant tumor, in any location of the body
10. Vaginal rejuvenation treatment, including laser treatments and radiofrequency therapy, within the 6 months prior to the Screening Visit
11. Subject has used the BTL EMSELLA device previously
12. Neurologic conditions deemed exclusionary by an investigator, including multiple sclerosis, spina bifida, Parkinson's, spinal cord injury, diabetic neuropathy etc.
13. Chronic pelvic pain > 4/10 VAS
14. Undiagnosed/unmanaged disorders of motility, including Irritable Bowel Syndrome (IBS)
15. Undiagnosed colorectal conditions
16. Bowel surgery in the past 12 months
17. Currently participating in an investigational study that may impact study results or previously received an investigational drug or treatment within 30 days of the Screening Visit
18. Current or history of any physical condition that, in the investigator's opinion, might put the subject at risk or interfere with study results interpretation

    * To preserve the integrity of the study, some criteria have been omitted. All criteria will be available to the public at the close of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
compare the efficacy of Emsella Chair to sham by evaluating the responder rate, where a subject is called a responder if there is ≥ 50% reduction from baseline in the number fecal incontinence episodes reported over 7 days on the bowel diary. | 4 weeks after completing all treatments
  Compare the efficacy of Emsella Chair to sham by evaluating the total number of fecal incontinence episodes reported in a bowel diary. Subjects will complete a 7 day bowel diary and record the number and consistency of bowel movements.

SECONDARY OUTCOMES:
Efficacy of Emsella chair vs. sham Emsella in relation to the change in quality of life (QoL) score as measured by the Cleveland Clinic Incontinence Score (Wexner). | 4 weeks after completing primary endpoint visit
  Compare the efficacy of the Emsella Chair versus sham in relation to the change in patient quality of life (QoL) score as measured by the Cleveland Clinic Incontinence score (Wexner). Subjects will report if their lifestyle is altered by incontinence, degree of occurrence is measured as 0 = never, 1 = rarely, 2 = sometimes, 3 = usually, 4 = always. High score = poor quality of life.
Efficacy of Emsella chair vs. sham Emsella in relation to the change in quality of life (QoL) score as measured by the Fecal Incontinence Quality of life scale (FIQOL). | 4 weeks after completing primary endpoint visit
  Compare the efficacy of the Emsella Chair versus sham in relation to the change in patient quality of life (QoL) score as measured by the FIQOL. Scales range from 1 to 4; with a 1 indicating a lower functional status of quality of life. Scales are divided into the following categories lifestyle, coping/behavior, depression/self perception, and embarrassment.
Efficacy of Emsella chair vs. sham Emsella in relation to the change in Fecal Incontinence severity as measured by the Cleveland Clinic Incontinence Score (Wexner). | 4 weeks after completing primary endpoint visit
  Compare the efficacy of the Emsella Chair versus sham in relation to the change in patient FI score as measured by the Cleveland Clinic Incontinence score (Wexner). The type of incontinence of stool (solid, liquid, gas, wears pad, lifestyle altered) are reported by the subject. Each question is measured as; 0 = never, 1 = rarely, 2 = sometimes, 3 = usually, 4 = always. The higher the score the more severe the condition.
Efficacy of Emsella chair vs. sham Emsella in relation to the change in self-reported impression of Fecal Incontinence severity. | 4 weeks after completing primary endpoint visit
  The change in self-reported impression of Fecal Incontinence severity as measured by the Patient Global Impression of Severity Scale (PGI-S). Subjects will check the box that describes how their condition is now. The available options are 1 =normal, 2 = mild, 3 = moderate, or 4 = severe. A higher score indicates a poorer outcome.
Efficacy of Emsella chair vs. sham Emsella in relation to the change in subject-reported impression of Fecal Incontinence improvement. | 4 weeks after completing all treatments
  The change in subject-reported impression of Fecal Incontinence improvement as measured by the Patient Global Impression of Improvement Scale (PGI-I). The subject will select one of the following options, (1 = very much better, 2 = much better, 3 = a little better, 4 = no change, 5 = a little worse, 6 = much worse, 7 = very much worse) to describe fecal incontinence symptoms now versus to prior to study treatment. A higher score indicates worsening of symptoms and poorer outcome.
Durability of this study to determine whether subjects in the Emsella Chair group continue to have a higher responder rate than the Sham group. | 4 weeks after completing all treatments
  Responders will be subjects that report positive outcomes (i.e. improvement in symptoms and decreased frequency of occurrence of symptoms) in the previously mentioned outcome measures.
Determine the safety and tolerability of the Emsella Chair versus sham through the incidence of Treatment-Emergent adverse events | 4 weeks after completing all treatments
  Safety and tolerability will be assessed in relation to the incidence of treatment- emergent adverse events reported.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Beaumont Hospital-Royal Oak
Locations (1):
- Beaumont Hospital-Royal Oak, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No